CLINICAL TRIAL: NCT01282489
Title: Evaluation of Methods to Asses Visual Prosthesis Systems Using Sighted Volunteers and Visual Reality Simulator
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Shamoon College of Engineering (Unknown)
Responsible Party: Sponsor
Other Study IDs: MMC11142-2010CTIL
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2014-06

CONDITIONS: Focus of Study: Finding Ways to Evaluate Visual Prosthesis Systems

SUMMARY:
A basic requirement for every therapeutic procedure is that there be an objective and validated method to assess the benefit of the treatment for the patient. Currently, there is no acceptable procedure to quantify the benefit obtained from visual prostheses.

The goal of the proposed research is to evaluate visual tasks and tests that will be given to a very large number of volunteers with normal vision who will be using a novel virtual prosthesis simulator. This device will simulate the realistic visual information that a visual implant can provide and will be used to measure implants in current clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Normal or corrected to normal sight (up to +/- 3.5 D) - Healthy Age 18 to 45

Exclusion Criteria:

Had any incident of dizziness from video or computer game Minors or special population

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers with normal or corrected to normal sight
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
quantitative comparison with standard visual acuity test (ETDRS) | December 1, 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Neurology, Meir Medical Center, Kfar Saba, Israel